CLINICAL TRIAL: NCT01854268
Title: Respiratory Kinematics During Voluntary and Reflex Cough in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 32-2013
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Cough
Keywords: cough
MeSH Terms: conditions — Cough | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy adults who receive capsaicin (Experimental): Single treatment consisting of healthy adults.
  Interventions: Drug: Healthy adults who receive capsaicin

INTERVENTIONS:
Drug: Healthy adults who receive capsaicin — Participants will be seated in a comfortable chair and fitted with cotton elastic bands designed to measure changes in chest wall and abdominal movement during cough. The participant will hold a facemask attached to a pneumotachograph, nebulized, and dosimeter. The participant will receive 3 nebulized doses of 200 microMolar capsaicin through the facemask. The participants will have a minute in between each presentation and water will be available at all times.
  Other Names: capsaicin

SUMMARY:
Cough is a defensive behavior that involves three stages. A large inspiratory phase, a compression phase where the vocal folds close and subglottal pressure is developed, and an expiratory phase. Cough serves to protect the upper and lower airways from material such as liquids, solids, or saliva, that have been aspirated. There are two types of cough: voluntary and reflex cough. Voluntary cough involves a cough to command. Reflex cough is a cough that is generated secondary to a stimulus in or near the airway. There has been some research regarding the differences between voluntary and reflex cough. However, no research has described the differences in airflow or movement pattern (kinematics) between the two types of cough. This study seeks to determine the respiratory kinematics and airflow differences between voluntary and reflex cough in healthy participants.

DETAILED DESCRIPTION:
As a participant, completion of this study will require the following:

Investigators will first place cotton elastic bands around your chest and abdomen so that measures of chest wall and abdominal movements can be measured. Then, tests of your breathing made from pulmonary function testing will be completed.

Investigators will then have you complete a maximum inspiration followed by a maximum expiration three times.

Investigators will ask you to produce a voluntary cough three times into a facemask which is attached to a computer.

Then the investigators will provide you with nebulized water (FOG) through the facemask for up to a minute three times. You will have a minute break in between each presentation.

Finally, the investigators will provide you with a nebulized dose of Capsaicin, which is derived from hot peppers, through the same facemask used in all of the above tasks. You will receive three doses of capsaicin and be provided with water at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18-80 years.
* Ability to provide informed consent.

Exclusion Criteria:

* No history of smoking within the last 5 years as this reduces the sensitivity to capsaicin
* No history of neurological disease (i.e. Parkinson's disease, stroke, traumatic brain injury, etc.)
* No known allergy to capsaicin
* No history of respiratory disease (i.e. asthma, chronic obstructive pulmonary disease, or respiratory infection within the last 5 weeks.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra E. Brandimore, M.A., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Dauer Hall, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adults Who Receive Capsaicin: Single treatment consisting of healthy adults.
  Healthy adults received capsaicin: Participants were seated in a comfortable chair and fitted with cotton elastic bands designed to measure changes in the chest wall and abdomen during cough. Participants breathed through a facemask attached to a pneumotachograph, nebulizer, and dosimeter. Participants received 3 nebulized doses of 200 microMolar capsaicin through the facemask. The participants rested for a minute in between each presentation and water was available at all times.
  Pulmonary function testing: Investigators placed cotton elastic bands around the chest and abdomen so that measures of chest wall and abdominal movements could be measured. Forced vital capacity and rest breathing was completed.
  Nebulized water (Fog): The investigators provided nebulized water (FOG) through the facemask for up to a minute three times. A minute break was allotted between each presentation.
Period: Overall Study
Arm/Group | Healthy Adults Who Receive Capsaicin
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were evaluated one time. Therefore baseline evaluations were the only measures completed.
Groups:
- Healthy Adults Who Receive Capsaicin: Single treatment consisting of healthy adults.
  Healthy adults who receive capsaicin: Participants were seated in a comfortable chair and fitted with cotton elastic bands designed to measure changes in chest wall and abdominal movement during cough. The participant breathed through a facemask attached to a pneumotachograph, nebulizer, and dosimeter. The participant received 3 nebulized doses of 200 microMolar capsaicin through the facemask. The participants had a minute in between each presentation and water was available at all times.
  Pulmonary function testing: Investigators will first place cotton elastic bands around your chest and abdomen so that measures of chest wall and abdominal movements can be measured. Forced vital capacity and rest breathing maneuvers were completed.
  Nebulized water (Fog): The investigators will provide you with nebulized water (FOG) through the facemask for up to a minute three times. A minute break in between each presentation.
Arm/Group | Healthy Adults Who Receive Capsaicin
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 25
Lung volume initiation [Mean (Standard Deviation); unit: %vital capacity, relative to EEL] — Lung volume initiation (LVI), termination (LVT), and excursion (LVE) measurements during voluntary and reflex cough: mean percent vital capacity difference relative to end-expiratory level (EEL). Significant lung volume differences between reflex and voluntary cough
  %vital capacity, relative to EEL | 23.3 (5.8)
Peak expiratory airflow rate [Mean (Standard Deviation); unit: Liters/second] | 6.058 (.56)
Urge-to-cough [Median (Standard Deviation); unit: units on a scale] | 7 (.32)

OUTCOME MEASURES:

1. Primary Outcome: Lung Volume Initiation
Description: Respiratory kinematic measure: lung volume initiation (LVI) Lung volume initiation is a measure of the volume of air in the lungs prior to a respiratory task.
Time Frame: 1 hour
Population: 25 healthy young volunteers participated in this study. The average age was 23 years and none had a history of respiratory or neurological disease.
Measure: Mean (Standard Deviation); unit: % Vital Capacity, relative to EEL
Arm/Group | Healthy Adults Who Receive Capsaicin
Number analyzed (Participants) | 25
% Vital Capacity, relative to EEL | 23.3 (5.7)

2. Secondary Outcome: Peak Expiratory Airflow Rate
Description: Airflow measures: Peak expiratory airflow rate Peak expiratory flow rate is a measure of the velocity of air expelled from the respiratory apparatus during cough. Measured in liters/second.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: Liters/second
Arm/Group | Healthy Adults Who Receive Capsaicin
Number analyzed (Participants) | 25
Liters/second
  PEFR - Voluntary Cough | 6.058 (.56)
  PEFR - Reflex Cough | 5.437 (.43)

3. Secondary Outcome: Urge-to-cough
Description: Urge-to-cough: A measure of respiratory sensation that rates the perceived magnitude of the need to cough on a Borg scale (0=no urge-to-cough; 10=maximal urge-to-cough).
Time Frame: 1 hour
Measure: Median (Standard Error); unit: units on a scale
Arm/Group | Healthy Adults Who Receive Capsaicin
Number analyzed (Participants) | 25
units on a scale | 6 (.4)

ADVERSE EVENTS:
Time Frame: All study participants were recruited during one month.
Description: There were no adverse events associated with this protocol.
Groups:
- Healthy Adults Who Receive Capsaicin: Single treatment consisting of healthy adults.
  Healthy adults received capsaicin: Participants were seated in a comfortable chair and fitted with cotton elastic bands designed to measure changes in chest wall and abdominal movement during cough. The participant breathed through a facemask attached to a pneumotachograph, nebulizer, and dosimeter. The participant received 3 nebulized doses of 200 microMolar capsaicin through the facemask. The participants had a minute in between each presentation and water will be available at all times.
Arm/Group | Healthy Adults Who Receive Capsaicin
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes